CLINICAL TRIAL: NCT05458661
Title: Feasibility Investigation of Biometry and Tomography Measurements in a Heterogeneous Patient Cohort (BioBase)
Brief Title: Feasibility Investigation of Biometry and Tomography Measurements in a Heterogeneous Patient Cohort
Acronym: BioBase
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B2101CI
Record Dates: First submitted 2022-04-05; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Cataract; Lens Opacities; Artificial Lens Implant; Corneal Astigmatism; Corneal Defect; Corneal Deformity
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Intervention Model Description: all suitable/eligible subjects will undergo a series of biometry measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- recruited patient population (Other)
  Interventions: Device: Clinical Prototype BioBase (SN 07 and SN 08)

INTERVENTIONS:
Device: Clinical Prototype BioBase (SN 07 and SN 08) — Scheimpflug- or OCT based corneal tomographers with the ability to measure anterior and posterior corneal curvature maps >6mm diameter and corneal pachymetry maps >6mm.
  Other Names: IOLMaster 700 Vs. 1.90 (Carl Zeiss Meditec AG, Göschwitzer Straße 51-52, 07745 Jena); Pentacam HR (Oculus Optikgeräte GmbH, Münchholzhäuser Straße 29, 35582 Wetzlar); MS-39 (bon Optic Vertriebsges. mbH, Stellmacherstraße 14, 23556 Lübeck)

SUMMARY:
The planned clinical investigation will be conducted to acquire raw data for the development of the algorithm. The data acquisition is intended to obtain first impressions of the potential performance of the changed hardware and software components and to confirm the safety profile assessed by risk analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 21 years of age and older
* Able and willing to make the required study visit
* Able and willing to provide consent and follow study instructions
* Patients must have understood and signed the informed consent

Exclusion Criteria:

* Any performed contact measurements or examinations in which the eye is touched on the same day prior to the investigation measurement
* Physical inability to be positioned at the study devices (e.g. torticollis, head tremor, injuries at forehead or chin, etc.)
* Principal Investigator's determination that the subject is not suitable due to other medical condition (reasons to be listed on eCRF)
* Known Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Data collection for algorithm development - Cornea to retina Scan | day 1
  - Cornea to retina Scan (all axial measurements) The data will be used within the Carl Zeiss Meditec R&D department to further develop the algorithm of this device to get a next generation biometry device with automated base.
Data collection for algorithm development - Corneal topography | day 1
  - Corneal topography (raw data and images) including keratometry The data will then be used within the Carl Zeiss Meditec R&D department to further develop the algorithm of this device to get a next generation biometry device with automated base.
Data collection for algorithm development - - Anterior-segment OCT data | day 1
  - Anterior-segment OCT data The data will be used within the Carl Zeiss Meditec R&D department to further develop the algorithm of this device to get a next generation biometry device with automated base.
Data collection for algorithm development - Extended retina-scan | day1
  - Extended retina-scan The data will be used within the Carl Zeiss Meditec R&D department to further develop the algorithm of this device to get a next generation biometry device with automated base.
Data collection for algorithm development - Reference pictures for markerless alignment of toric IOL (sclera images) | day 1
  - Reference pictures for markerless alignment of toric IOL (sclera images) The data will be used within the Carl Zeiss Meditec R&D department to further develop the algorithm of this device to get a next generation biometry device with automated base.
Data collection for algorithm development - White-to-white determination | day 1
  - White-to-white determination The data will then be used within the Carl Zeiss Meditec R&D department to further develop the algorithm of this device to get a next generation biometry device with automated base.
Data collection for algorithm development - IOL Imaging pictures | day 1
  - IOL Imaging pictures The data will then be used within the Carl Zeiss Meditec R&D department to further develop the algorithm of this device to get a next generation biometry device with automated base.
Affected measurements - OCT measurements | day 1
  It will be investigated, whether the measurements with the study prototype device are affected by the base movement.
  - OCT measurements This outcome will be investigated by comparing the raw data of the study prototype device with the data measured with the marketed IOLMaster 700 and Pentacam / MS-39 devices.
  Non-optimal positioning and movement could possibly cause blurred images that would prevent a detailed analysis
Affected measurements - Keratometry and Topography measurements | day 1
  It will be investigated, whether the measurements with the study prototype device are affected by the base movement.
  - Keratometry and Topography measurements This outcome will be investigated by comparing the raw data of the study prototype device with the data measured with the marketed IOLMaster 700 and Pentacam / MS-39 devices.
  Non-optimal positioning and movement could possibly cause blurred images that would prevent a detailed analysis
Affected measurements - - WTW measurements | day 1
  It will be investigated, whether the measurements with the study prototype device are affected by the base movement.
  - WTW measurements This outcome will be investigated by comparing the raw data of the study prototype device with the data measured with the marketed IOLMaster 700 and Pentacam / MS-39 devices.
  Non-optimal positioning and movement could possibly cause blurred images that would prevent a detailed analysis

IPD SHARING:
Plan to Share IPD: No
no publications planned